CLINICAL TRIAL: NCT02172846
Title: A Phase I Study of Radiation Dose Intensification With Accelerated Hypofractionated Proton Therapy and Chemotherapy for Non-small Cell Lung Cancer
Brief Title: Hypofractionated Proton Beam Radiation Therapy, Paclitaxel, and Carboplatin in Treating Patients With Stage II-III Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201404047
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Proton Therapy; Paclitaxel; Albumin-Bound Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (PBT, paclitaxel, and carboplatin) (Experimental): CHEMORADIATION THERAPY:
  * PBT daily 5 days a week over 3 weeks for a total of 15 fractions
  * Paclitaxel intravenously (IV) over 1 hour weekly for 3 weeks
  * Carboplatin intravenously (IV) over 30 minutes weekly for 3 weeks.
  CONSOLIDATION CHEMOTHERAPY (B=beginning 4-6 weeks after completion of radiation therapy, patients may receive):
  * Paclitaxel IV over 1 hour on day 1
  * Carboplatin IV over 30 minutes on day 1
  * At the discretion of the treating physician
  * Treatment repeats every 3 weeks for 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: Proton beam radiation therapy (PBT); Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Radiation: Proton beam radiation therapy (PBT)
Drug: Paclitaxel
  Other Names: Abraxane®; Onxol®; Taxol®
Drug: Carboplatin
  Other Names: Paraplatin®; CBDCA

SUMMARY:
This phase I trial studies the side effects and best dose of hypofractionated proton beam radiation therapy when given together with paclitaxel and carboplatin in treating patients with stage II-III non-small cell lung cancer. Proton beam radiation therapy is a type of radiation therapy that uses streams of protons (tiny particles with a positive charge) to kill tumor cells. Giving proton beam radiation therapy at higher doses over fewer days (hypofractionation) may improve local control of the tumor. Giving hypofractionated proton beam radiation therapy with chemotherapy may be a better treatment for non-small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically proven diagnosis of non-small cell lung cancer.
2. Clinical AJCC stage II-III (AJCC, 7th ed.) with plans to be treated with concurrent chemoradiotherapy.

   1. Recurrent non-small cell lung cancer is allowed, provided the intent of the current treatment is curative and there has been no prior radiation to the thorax.
   2. Prior chemotherapy, immunotherapy, or targeted therapy is permitted as long as patients have recovered from prior toxicities to grade ≤ 1
3. Appropriate stage for protocol entry based upon the following minimum diagnostic workup:

   1. History/physical examination within 30 days prior to registration;
   2. FDG-PET/CT scan for staging within 60 days prior to registration;
   3. MRI scan with contrast of the brain (preferred) or CT scan of the brain with contrast within 60 days prior to registration.
4. Zubrod Performance Status 0-2 within 30 days prior to registration.
5. Age ≥ 18 years.
6. CBC/differential obtained within 30 days prior to registration, with adequate bone marrow function defined as follows:

   1. Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3;
   2. Platelets ≥ 100,000 cells/mm3;
   3. Hemoglobin ≥ 8.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable.);
7. AST and ALT ≤ 1.5 upper limit of normal within 30 days prior to registration.
8. Total bilirubin ≤ 1.5 upper limit of normal within 30 days prior to registration.
9. Serum creatinine < 1.5 mg/dL or calculated creatinine clearance ≥ 50 mL/min within 30 days prior to registration estimated by the Cockcroft-Gault formula:

   Creatinine Clearance (male) = [(140 - age) x (wt in kg)] [(Serum Creatinine mg/dl) x (72)]

   Creatinine Clearance (female) = 0.85 x Creatinine Clearance (male)
10. Peripheral neuropathy ≤ grade 1 at the time of registration.
11. Presence of measurable or evaluable disease.
12. Negative serum or urine pregnancy test within 2 weeks prior to registration for women of childbearing potential.
13. Women of childbearing potential and male participants must agree to use a medically effective means of birth control throughout their participation in the treatment phase of the study.
14. Able to understand and willing to sign an IRB-approved informed consent document.

Exclusion Criteria:

1. Severe, active comorbidity, defined as follows:

   1. Unstable angina, history of myocardial infarction and/or congestive heart failure requiring hospitalization within the last 6 months;
   2. Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration;
   3. Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration;
   4. Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol;
   5. Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive. Protocol-specific requirements may also exclude immuno-compromised patients.
2. Prior radiotherapy to the thorax.
3. Currently receiving any other investigational agents.
4. Pregnant or breastfeeding.
5. Presence of a cardiac pacemaker (due to the risk created by the proton magnet).

Inclusion of Women and Minorities

Both men and women and members of all races and ethnic groups are eligible for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-05-22 (Actual); Primary Completion 2016-08-23 (Actual); Study Completion 2017-10-02 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of hypofractionated proton beam therapy (PBT) with chemotherapy | Up to 6 months
  Common Terminology Criteria for Adverse Events version 4 (CTCAE) will be used. The MTD will be chosen as the dose that yields a posterior estimate of toxicity closest to 20% while being between 15% and 25%.
  Dose limiting toxicity will be defined as toxicity that occurs within 6 months from the start of treatment, is possibly, probably or definitely related to treatment, and is related to the following
  Grade 3-5 pericardial effusion, pericarditis, restrictive cardiomyopathy, hemorrhage (pulmonary or upper respiratory), excluding nose, larynx, or pharynx, brachial plexopathy, laryngeal nerve dysfunction, myelitis, phrenic nerve dysfunction , atelectasis (grade 4-5 only), pulmonary fistula, hypoxia (provided grade 3 is worse than baseline), obstruction/stenosis of the airway, pleural effusion, pneumonitis, pulmonary fibrosis Grade 4-5 dysphagia, esophagitis, esophageal fistula, obstruction, perforation, stricture/stenosis, ulcer, and hemorrhage Grade 4-5 skin Any grade 5

SECONDARY OUTCOMES:
Incidence of acute toxicities | Up to 6 months
  Common Terminology Criteria for Adverse Events version 4 (CTCAE) will be used.
  Adverse events will be tabulated by type and grade.
Incidence of late toxicities as defined | Up to 1 year
  Common Terminology Criteria for Adverse Events version 4 (CTCAE) will be used.
  Adverse events will be tabulated by type and grade.

CONTACTS AND LOCATIONS:
Overall Officials: Cliff Robinson, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu